CLINICAL TRIAL: NCT04185077
Title: The Efficiency and Safety of Bivalirudin in latE percuTaneous Coronary inTervention for Patients With ST-Elevation Myocardial InfaRction (BETTER Trial)
Brief Title: Bivalirudin in Late PCI for Oatients With STEMI
Acronym: BETTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Shenghua Zhou, Director, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJUHFCSOARF201901-20
Record Dates: First submitted 2019-11-29; First posted 2019-12-04 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: STEMI; late PCI; Bivalirudin; anticoagulation
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — bivalirudin; Antithrombins; Heparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Bivalirudin (Salubris Pharmaceuticals Co) was given as a bolus of 0.75mg/kg followed by infusion of 1.75mg/kg/h during the PCI procedure and for at least 30 minutes but no more than 4 hours afterwards. Following this mandatory infusion, a reduced-dose infusion (0.2mg/kg/h) for up to 20 hours could be administered at physician discretion. An additional bivalirudin bolus of0.3mg/kgwasgivenif the activatedclotting time 5minutes after the initial bolus (measuredwith the Hemotec assay) was less than 225 seconds.
  Interventions: Drug: Bivalirudin
- Control (Active Comparator): a bolus dose of 100 U/kg Heparin was administered according to current guidelines.Additional heparinwasadministered if the post-bolus activated clotting time was less than 225 seconds.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Bivalirudin — Bivalirudin (Salubris Pharmaceuticals Co) was given as a bolus of 0.75mg/kg followed by infusion of 1.75mg/kg/h during the PCI procedure and for at least 30 minutes but no more than 4 hours afterwards. Following this mandatory infusion, a reduced-dose infusion (0.2mg/kg/h) for up to 20 hours could be administered at physician discretion. An additional bivalirudin bolus of0.3mg/kgwasgivenif the activatedclotting time 5minutes after the initial bolus (measuredwith the Hemotec assay) was less than 225 seconds.
  Other Names: Direct thrombin inhibitor
  Arms: Experimental
Drug: Heparin — a bolus dose of 100 U/kg was administered according to current guidelines.Additional heparinwasadministered if the post-bolus activated clotting time was less than 225 seconds.
  Other Names: unfractionated heparin
  Arms: Control

SUMMARY:
Bivalirudin is recomended by guidelines during primary PCI procedure for patients with STEMI. However, there is a large number of STEMI patients who missed the primary PCI. So the investigators aim to study the efficiency and safety of bivalirudin as the anticoagulation therapy during late PCI.

DETAILED DESCRIPTION:
Antithrombotic therapy is essential to prevent adverse ischemic events, especially stent thrombosis and reinfarction during and after primary percutaneous coronary intervention (PCI) in patients with acute myocardial infarction (AMI). Bivalirudin is emerging as an alternative for heparin during PCI procedure1.

Bivalirudin (BIV) a synthetic, bivalent, 20-amino acid direct thrombin inhibitor, was found to have the advantages of inhibiting fibrin-bound thrombin, a predictable effect of anticoagulation, and a short half-life of approximately 30 minutes in humans with normal renal function. BIV has been introduced in percutaneous coronary interventions (PCIs) especially for patients with ACS. Compared with heparin, series clinical trials indicated that BIV was not inferior to UFH as a procedural anticoagulant and there was no increased bleeding.

In the real world, there are as many as 47.1% patients with STEMI can not get early reperfusion therapy. Huge number of patients missed the best time window for PCI. For these patients, the usual PCI procedure are usually performed 1-2 weeks after attack, which is called late PCI.

For patients with STEMI, Bivalirudin is recomended by guidelines in ESC during PCI procedure. However, the evidences (ACUITY，HORIZONS-AMI，EUROMAX, EAT-PPCI，BRIGHT, VALIDATE-SWEDEHEART) supporting the guideline nearly all comes from primary PCI for STEMI, which means there has no clinical trials focus on late PCI for patients with STEMI yet.

Clinically, late PCI, defined as the time to open an infarct-related artery (IRA) from symptoms onset > 7 days (when the myocardial condition is considered stable), is practiced commonly for these late presenters. Whether late PCI is adequately beneficial is controversial. Currently, heparin is applied during late PCI as the anticoagulation therapy, it is still unknown of the efficiency and safety for bivalirudin as the anticoagulation therapy during late PCI.

So in this RCTs, the investigators aim to study the efficiency and safety of bivalirudin as the anticoagulation therapy during late PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years.
2. Patients with ST-segment elevation MI (STEMI) undergoing late PCI 24 hours to 2 weeks after symptom onset. STEMI was defined as ST-segment elevation ≥0.1 mV in ≥2 contiguous leads or documented newly developed left bundle branch block.
3. Patients with develop Q-waves at presentation and with clear culprit vessel confirmed by angiography or other clinical evidences.
4. No any other anticoagulation therapy 12 hours before late PCI.

Exclusion Criteria:

- STEMI patients undergoing primary PCI in 24 hours after symptom attack; patient unwilling or unable to provide written informed consent. thrombolytic therapy administered before randomization; any condition making PCI unsuitable or that might interfere with study adherence;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-11-30 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of net adverse clinical events | 30 days after discharge
  a composite of major adverse cardiac or cerebral events (all-cause death, reinfarction, ischemia-driven target vessel revascularization, or stroke) or any bleeding as defined by the Bleeding Academic Research Consortium(BARC) definition (grades 1-5).

SECONDARY OUTCOMES:
Rate of major adverse cardiac or cerebral events | 30 days after enrollment
  all-cause death, reinfarction, ischemia-driven target vessel revascularization, or stroke
Rate of any bleeding | 30 days after enrollment
  Bleeding was considered medically actionable if BARC types 2 through 5 and was considered major if BARC types 3 through 5 occurred.
Rate of stent thrombosis | 30 days after enrollment
  according to the Academic Research Consortium criteria
Rate of acquired thrombocytopenia | 30 days after enrollment
  defined as a platelet count decrease ofmore than50%or more than 150 × 109/L frombaseline